CLINICAL TRIAL: NCT01728532
Title: Open, Randomized Multicentric Trial Evaluating the Efficacy and the Clinical Tolerance of PA0903 as Root Canal Sealer
Brief Title: Open, Multicentric Trial Evaluating the Efficacy and the Clinical Tolerance of PA0903 as Root Canal Sealer
Acronym: PA0903
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascopharm Groupe Novasco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/001
Record Dates: First submitted 2012-11-06; First posted 2012-11-20 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Root Canal Obturation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulp Canal Sealer (Kerr) (Active Comparator): zinc oxide eugenol sealer
  Interventions: Device: Pulp Canal Sealer (Kerr)
- PA0903 (Experimental): type C implant according to ISO 7405:2008 and ISO 10993 guidelines.
  Interventions: Device: PA0903

INTERVENTIONS:
Device: Pulp Canal Sealer (Kerr) — permanent obturation of the root canal space with the aid of obturating points
  Arms: Pulp Canal Sealer (Kerr)
Device: PA0903 — Sealing performed by the dentist , coronal obturation placed after the canal obturation
  Arms: PA0903

SUMMARY:
TRIAL TITLE: Open, randomized multicentric trial evaluating the efficacy and the clinical tolerance of PA0903 as root canal sealer

SPONSOR:

SEPTODONT, 58 rue du Pont de Créteil, 94107 Saint Maur des Fossés cedex Tel : + 33 1-49-76-74-26, Fax. : + 33 1- 49-76-71-91

Reference protocol: 11/001

PRODUCT NAME: PA0903

MEDICAL DEVICE:

Class III: Root canal sealer Dose: not applicable Application : one single time

DEVELOPMENTAL PHASE: not applicable (medical device class III)

DETAILED DESCRIPTION:
METHODOLOGY:

This study is performed only in adults who required a non-surgical root canal obturation. The studied indication is the root canal sealing.

This multi-centre and open-label study comprises two groups corresponding to tested root canal sealer (a reference product and investigational product). Randomization is required.

Investigational product that is a dental cement based on biosilicate technology (PA0903) will be applied with lateral compaction or single cone technique. On the contrary, reference product that is a zinc oxide-eugenol used in dental practice (Pulp Canal Sealer) will be applied with a single wave technique.

Study start: 01/12/11

Inclusion period: 24 months

Study duration: 2 years after the end of inclusion period

OBJECTIVES: The trial objective is to illustrate the clinical and radiographic outcome of PA0903 in the described indication.

Primary objectives:

The primary objective is to evaluate: clinical and radiographic outcome of root canal treatment at two years when using PA0903 as an endodontic sealer with gutta-percha. The success rate is defined as no pain (score of 0 at the VAS scale) and absence or decrease in the size of LEO (fulfilment of Strindberg's criteria). If a pre-existing lesion, the size decrease associated with normal contours, width and structure of the periodontal margines is considered as success. All cases in which lesion increases or is stabilized after 2 years were judged as unsuccessful . Moreover, all cases in which Strindberg's criteria if they are suitable were not fulfilled were judged as unsuccessful. A follow-up of two years is described as the predictive time of success.

Secondary objective:

The secondary objectives are to evaluate the following criteria and in an indicative way, to compare them between patients receiving the PA0903 and those receiving the reference product:

- The success rate at each time point and also the components of this composite variable (i.e. pain and Healing process for total class (vital teeth and necrotic teeth) of endodontic status of teeth).

In case of pre-existing LEO associated with necrotic teeth, size of LEO and suitable Strindgberg's criteria will be used to judge the outcomes of the root canal therapy as described below :

At visit 2 (6 months) treatment is considered successful when LEO is stable or decreased in comparison with V0 associated with Strindberg's criteria suitable.

At V3 (1 year), treatment is considered successful when LEO is decreased in comparison with V2 associated with Strindberg's criteria suitable.

* the Healing process associated with PA0903 application in each endodontic status
* the handling, consistency and physical characteristics of PA0903
* the longevity and safety of the product associated with PA0903 after two years.

TRIAL POPULATION AND NUMBER OF PATIENTS: about 60 patients will have to be included in the study, 20 by center with a ratio 2 (PA0903): 1 (reference). Adults will be included without gender distinction.

Coordinating center Endodotontic service of Pitié Salpétrière Pitié Salpétrière Hospital 75634 Paris Cedex 13 France

DURATION OF TREATMENT:

The product is applied on D0 (inclusion) of the study. The follow-up period includes 2 years with 4 visits: Visit 1(Week 2), Visit 2 (Month 6), Visit 3 (Year 1) and Visit 4 (Year 2).

ELIGIBILITY:
Inclusion Criteria

* Male or female >18 years old
* provide signed, informed consent.
* be affiliated to social security.

In addition, the subjects must fulfill all of the following criteria for root canal sealer treatment:

* Permanent mature single rooted teeth : maxillary incisors, mandibular incisor with only one canal, upper and lower canine, upper and lower premolars with only one canal
* Permanent mature mandibular molars Pulp status
* Vital pulp that needs pulpectomy without clinical and/or radiological findings of apical periodontitis.
* Irreversible pulpitis with or without pain
* Non infected tooth that positively responds of pulp vitality test Or necrotic pulp with and without radiographic signs of apical pathosis Periodontal status
* No active periodontal disease

Exclusion criteria:

* History of malignancy in the last 5 years.
* Systemic disease not stabilized within 1 month before the Inclusion Visit (e.g., diabetes, thyroid malfunction, uncontrolled autoimmune disease) or judged by the investigator to be incompatible with the study (e.g. current systemic infections) or condition incompatible with the frequent assessments needed by the study.
* Risk A cardiopathies
* Known hypersensitivity to one of the components of the study or procedural medications.
* Presence or history of severe systemic allergy.
* Presence or history of drug addiction or alcohol abuse.
* Patient who has participated in a clinical trial with a new active substance during the month before study entry.
* Participation in another clinical study at the same time as the present study.
* Known pregnancy or lactation at study entry.
* Patients with legal protection

Specific criteria relative to root canal sealing are:

* Extreme curvature of the canals
* Dilacerations
* Root dilacerations and sharp apical curvature for mandibular molars
* Superimposition of mesial canals for mandibular molar
* Large peri-apical radiolucencies
* Periodontal disease
* Not primary endodontic treatment
* Perforated root canals
* Supracrestal iatrogenic perforation
* Inadequate or insufficient periodontal support
* Combined endo-periodontal lesion
* Loss of tooth structure (Coronal decay and/or concomitant root decay) compromising the tooth's maintenance on the dental arch)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
clinical and radiographic outcome of PA0903 as root canal sealer | 2 years
  to evaluate clinical and radiographic outcome of root canal treatment at two years when using PA0903 as an endodontic sealer with gutta-percha. The success rate is defined as no pain (score of 0 at the VAS scale) and absence or decrease in the size of LEO (fulfilment of Strindberg's criteria). If a pre-existing lesion, the size decrease associated with normal contours, width and structure of the periodontal margines is considered as success. All cases in which lesion increases or is stabilized after 2 years were judged as unsuccessful .A follow-up of two years is described as the predictive time of success.

SECONDARY OUTCOMES:
Secondary outcomes | 2 years
  - The success rate at each time point and also the components of this composite variable (i.e. pain and Healing process for total class (vital teeth and necrotic teeth) of endodontic status of teeth).
  In case of pre-existing LEO associated with necrotic teeth, size of LEO and suitable Strindgberg's criteria will be used to judge the outcomes of the root canal therapy as described below :
  At visit 2 (6 months) treatment is considered successful when LEO is stable or decreased in comparison with V0 associated with Strindberg's criteria suitable.
  At V3 (1 year), treatment is considered successful when LEO is decreased in comparison with V2 associated with Strindberg's criteria suitable.
  * the Healing process associated with PA0903 application in each endodontic status
  * the handling, consistency and physical characteristics of PA0903
  * the longevity and safety of the product associated with PA0903 after two years.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Simon, PhD, Principal Investigator — Hôpital Pitié Salpetrière, Paris, France
Locations (3):
- France (2):
  - Cabinet dentaire privé - 21, rue Fabre d'Églantine, Paris
  - Service d'endodontie de la Pitié Salpêtrière Hôpital de la Pitié Salpêtrière, Paris
- School of Dentistry Cardiff University, Cardiff, United Kingdom